CLINICAL TRIAL: NCT03925571
Title: Evaluation of the Effectiveness of Musicotherapy in Reducing Peroperative Anxiety and Post-surgical Pain in Dental Care
Brief Title: Musicotherapy in Reducing Peroperative Anxiety and Post-surgical Pain in Dental Care
Acronym: MUSANX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC17_0289
Record Dates: First submitted 2019-04-08; First posted 2019-04-24 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Dental Pain and Sensation Disorders
MeSH Terms: conditions — Toothache; Sensation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music-listening group (Experimental): patient will listen to music during the dental surgery (1 to 1h30 hours).
  Interventions: Other: musicotherapy
- non music-listening group (No Intervention): patient will receive their dental intervention without music-listening.

INTERVENTIONS:
Other: musicotherapy — If the patient is randomized in the experimental group, he listens the Music-care® playlists and chose two closed to his musical tastes. The playlists are unique compositions create by Music-care® (french company), not known from the general public, categorized by theme (jazz, rock, world music…).
  Arms: music-listening group

SUMMARY:
The main purpose of MUSANX study is to highlight analgesic effectiveness of musicotherapy in post-surgical periodontal and implant; and to measure its per-operative anxiolytic effectiveness

DETAILED DESCRIPTION:
This study will be on music use as musicotherapy "receptive " or " passive ", using hearing aid for listening in order to relax and reduce the anxiety and pain state of the patient. This care will be focused on the acute stress and pain during the dental care.

Another major secondary purpose will consist to explore the anxiolytic effect of the musicotherapy on diverse stress markers such as heart rate, respiratory rate, salivary cortisol ratio and electro-dermal intensity (RED).

ELIGIBILITY:
Inclusion Criteria:

* Majors aged between 18 and 55 years, with an appropriate hearing and able to use Music-Care© (selection of the playlist via internet access),
* Needing treatment in odontology - periodontal surgery (coronary elongation or sanitation surgery or muco-gingival surgery) or implantary surgery (placement of an unit implant or two implant in the same localization),
* Oral and dated consent,
* Agreeing to be contacted via phone at J+1 and to fill follow-up study documents,
* Profiting of social security or CMU.

Exclusion Criteria:

* Patients with a long-term taking of anxiolytic or analgesic,
* Regular consumer of soft drug (cannabis) or hard drug (opioid),
* Patient with medical history of psychiatry (mental harm), hearing problem, cognitive and behavioural impairment (claustrophobia), sensory disabilities,
* Patient with problems of hemostasis,
* Majors under trusteeship or guardianship,
* Pregnant women or lactating,
* Minors,
* Protected person, deprived of freedom or under justice safeguard,
* Profiting of a medical help from government (AME),
* Not contactable after care,
* Patient with hepatic impairment,
* Patient with dry mouth,
* Patient relevant a suboptimal hearing incompatible with musicotherapy or inability to use Music-care®.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 24 hours after the dental surgery
  the pain intensity will be measured with the Visual analogue scale (VAS).

SECONDARY OUTCOMES:
Efficacy of musicotherapy | 24, 48 and 72 hours
  Evaluate the anxiolytic effectiveness of " passive " musicotherapy on the reduction of peroperative anxiety during the dental surgery by STAY questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Assem Soueidan, Pr, Study Chair — Nantes University Hospital; Olivier Bonnot, Pr, Study Director — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided